CLINICAL TRIAL: NCT07363096
Title: Comparison Of Single- Versus Two-Level Erector Spinae Plane Block For Postoperative Analgesia In Patients Undergoing Lumbar Stabilization Surgery
Brief Title: Single- Versus Two-Level ESP Block for Analgesia After Lumbar Stabilization Surgery
Acronym: ESP-Lumbar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Hatice Ayça Sarıbudak, Anesthesiology and Reanimation Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2023-250
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management; Lumbar Spinal Fusion Surgery; Erector Spina Plan Block
Keywords: Erector Spina Plane Block; Acute Pain; Postoperative Pain Management
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Level Erector Spinae Plane Block (Active Comparator): Participants in this arm will receive an ultrasound-guided erector spinae plane (ESP) block performed at a single vertebral level corresponding to the surgical site, in addition to standardized general anesthesia and postoperative multimodal analgesia.
  Interventions: Procedure: Single-Level Erector Spinae Plane Block
- Two Level Erector Spinae Plane Block (Active Comparator): Participants in this arm will receive an ultrasound-guided erector spinae plane (ESP) block performed at two adjacent vertebral levels, in addition to standardized general anesthesia and postoperative multimodal analgesia.
  Interventions: Procedure: Two-Level Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Single-Level Erector Spinae Plane Block — Ultrasound-guided erector spinae plane block performed at a single vertebral level for postoperative analgesia.
  Arms: Single Level Erector Spinae Plane Block
Procedure: Two-Level Erector Spinae Plane Block — Ultrasound-guided erector spinae plane block performed at two adjacent vertebral levels for postoperative analgesia.
  Arms: Two Level Erector Spinae Plane Block

SUMMARY:
Lumbar stabilization surgery is commonly associated with moderate to severe postoperative pain. Effective pain control is important to improve patient comfort, early mobilization, and recovery. The erector spinae plane (ESP) block is a regional anesthesia technique that has been increasingly used for postoperative pain management in spine surgery.

This study aims to compare the effectiveness of single-level versus two-level ultrasound-guided ESP block for postoperative pain control in patients undergoing lumbar stabilization surgery. Patients will be randomly assigned to receive either a single-level ESP block or a two-level ESP block in addition to standard analgesic treatment.

Postoperative pain scores, opioid consumption, and the incidence of side effects will be evaluated during the postoperative period. The results of this study may help determine the most effective ESP block technique for pain management after lumbar stabilization surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III,
* BMI:18-40,
* Patients undergoing lumbar stabilization surgery involving 2 to 4 vertebral levels
* Patients who personally provide written informed consent to participate in the study

Exclusion Criteria:

* Patients with chronic pain conditions
* Patients with a history of chronic opioid use
* Patients undergoing emergency lumbar stabilization surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Remifentanyl Consumption | During the intraoperative period
  The amount of Remifentanyl that patients need to maintain anesthesia during the intraoperative period will be recorded

SECONDARY OUTCOMES:
Pain Scores | First 24 hours after surgery
  Pain will be assessed at rest and while movement using the from 0 ( no pain) to 10 (worst pain). Pain assessment will be done at the 1st, 2nd, 4th, 12th and 24th hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No